CLINICAL TRIAL: NCT03335930
Title: Tri-Service General Hospital, National Defense Medical Center
Brief Title: Exercise-induced Blood Glucose Response in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, CHIA-HUEI LIN, PhD, Assistant Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TSGHIRB: 097-05-157
Record Dates: First submitted 2017-11-05; First posted 2017-11-08 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: exercise; blood glucose response; metabolic control; type 2 diabetes.
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: 1. Participants were randomly assigned to one of three exercise times (morning/08:00-10:00, afternoon/14:00-16:00 evening/18:00-20:00).
  2. Training protocol: Treadmills were used for the aerobic exercise training. Participants received supervised exercise training three times per week on alternate days for 12 weeks at the medical centre.
  3. All participants followed this training protocol and maintained their usual lifestyles. The duration of each training session was 30 minutes and took place 1 to 2 hours after a meal.
  4. The intensity of the training was set at 60% VO2max (approximately equal to 72% HRmax) obtained from the GXT.
  5. During each session of the 30-minute aerobic exercise training, the patient's heart rate was maintained at 72% of heart rate maximal on treadmill. Appropriate speed and grade were used to achieve the target heart rate being tracked by the heart rate monitor and to accurately control the required exercise intensity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Morning exercise (Experimental): To exercise at morning (08:00-10:00)
  Interventions: Behavioral: a 12-week moderate-intensity exercise training
- Afternoon exercise (Active Comparator): To exercise at afternoon (14:00-16:00)
  Interventions: Behavioral: a 12-week moderate-intensity exercise training
- Evening exercise (Active Comparator): To exercise at evening (18:00-20:00)
  Interventions: Behavioral: a 12-week moderate-intensity exercise training

INTERVENTIONS:
Behavioral: a 12-week moderate-intensity exercise training — a 12-week, aerobic, moderate-intensity exercise training
  Other Names: aerobic exercise training

SUMMARY:
Exercise is recommended for type 2 diabetes, which is a global health problem. However, during a moderate-intensity exercise training there is an unpredictable risk of hypoglycemia for patients with type 2 diabetes. Therefore, the investigators aim to explore trends in blood glucose levels in response to a 12-week moderate-intensity exercise training in patients with type 2 diabetes and to explore the predictors of post-exercise blood glucose (PEBG) and exercise-induced glucose response (EIGR). A descriptive and longitudinal design was conducted. Eligible type 2 diabetes patients were recruited from outpatient clinics of a medical center in Taiwan and invited to participate in a 12-week moderate-intensity exercise-training program. Each participant received 36 repeated measures of blood glucose during the exercise training program. Participants were randomly assigned to one of three exercise times (morning/afternoon/evening). Each exercise session was took place 1 to 2 hours after a meal. Capillary blood glucose levels were measured pre- and post-exercise. The EIGR was calculated from subtracting the PEBG from the before-exercise blood glucose (BEBG). Generalized estimating equation was used to examine the trends and predictors of PEBG and EIGR.

DETAILED DESCRIPTION:
A prospective and longitudinal design using purposive sampling was used. All eligible Taiwanese participants with T2DM at a medical centre were invited to participate in the exercise-training programme that included three sessions per week, 30 minutes per session for 12 weeks (total 36 sessions). Each participant's exercise sessions were equally randomised into three times of day (morning/08:00-10:00, afternoon/14:00-16:00 evening/18:00-20:00) using permuted-block randomisation. Capillary blood glucose samples were obtained before and after each 30-minute moderate-intensity (60% VO2max) exercise session. The EIGR, described as the difference between BEBG and PEBG values, was calculated.

Participants and setting: Participants with T2DM being seen at an outpatient clinic in a northern Taiwan medical centre were recruited by an endocrinology/metabolism physician. Participants, 40-60 years of age, diagnosed as having T2DM based on the criterion of the American Diabetes Association, and were being treated with oral antidiabetic medications only were eligible. Other inclusion criteria were (1) able to speak and understand Mandarin; (2) able to walk without assistance; (3) have no regular exercise habit; and (4) agree to join in a 12-week moderate-intensity exercise training after passing a graded exercise test (GXT), described below. Exclusion criteria included insulin therapy, a history of cancer, end-stage renal disease with dialysis, an inability to participate in exercise training due to comorbid neurological and musculoskeletal conditions, severe comorbidity or complications such as heart failure, autonomic neuropathy, and recent stroke within 6 months.

Under an effect size of 0.2, thirty-six numbers of measurements with a correlation efficient of 0.32 among repeated measures, an expected power of 0.7 to 0.8, and an alpha of 0.05, the required sample size was between 12 and 14 based on repeat measures (within factors). Therefore, initially 52 T2DM patients were approached and seventeen eligible participants were invited by a research nurse to receive GXT. Fifteen passed the exercise test based on the guidelines of the American College of Sports Medicine (ACSM) for exercise testing. A second research nurse assessed the baseline characteristics (eg, self-reported demographics and lifestyle patterns, blood analyses and anthropometric measures) of the final 15 participants. Participants were then invited to perform 36 exercise sessions (3 sessions/week for 12 weeks), which were randomly assigned to morning, afternoon, or evening using permuted-block randomization, except two dropped out after exercise test.

Graded exercise test: The GXT was performed using a motorised treadmill (Trackmaster 400, JAS Fitness System, USA) for identification of maximum oxygen uptake (VO2max), maximum heart rate (HRmax) and the risk for potentially life-threatening cardiovascular disease (eg, myocardial infarction). GXT procedures followed a modified Balke protocol.20 Two observers (a medical/rehabilitation doctor and a research nurse) were involved with each patient throughout the GXT. The GXT was immediately stopped if the patient complained of exhaustion; reached maximum heart rate or VO2max, determined by the maximal amount of blood the heart pumps per minute (cardiac output) and the amount of oxygen utilised by the exercising muscles (arterial-venous oxygen difference); had a respiratory exchange ratio >1.15; developed symptoms such as chest pain, dyspnea, pallor, diaphoresis or dizziness; had systolic pressure greater than 250 mm Hg or diastolic pressure greater than 120 mm Hg; had a decrease in systolic pressure of more than 10 mm Hg compared to the systolic pressure at rest; or requested stopping the test.

Ethical consideration: Institutional review board approval (TSGHIRB: 097-05-157) was obtained from Tri-Service General Hospital in Taiwan. All participants gave written informed consent when invited to join the study. Participants were assured that their participation was entirely voluntary and that they could withdraw at any time.

Data analysis: Statistical analyses were performed by SPSS version 16.0 (SPSS Inc., Chicago, IL). Descriptive data are presented as mean/standard deviation (SD) and numbers/percentage (%). Before evaluating the trend of blood glucose response during the 12-week/36-session exercise-training programme, two variables including "training month (1st, 2nd and 3rd month of the training)" and "timing of exercise sessions (1st to 36th session of exercise)" were coded. With generalised estimating equations (GEE), the investigators examined the change patterns of BEBG, PEBG and EIGR over time during the training programme. The trend analyes of BEBG, PEBG and EIGR were adjusted for covariates (i.e, age, gender, baseline body mass index, VO2max, HgbA1c, antidiabetic medication (metformin, sulfonylureas or repaglinide) and exercise time of day (morning, afternoon or evening). When evaluating the predictors of EIGR and PEBG, univariable analysis was applied first and, following the multivariable analysis, incorporated with those significant covariates from univariable analysis. All of the statistical analyses were two-tailed and considered significant at p < .05.

ELIGIBILITY:
Inclusion Criteria:

* 40-60 years of age
* diagnosed as having T2DM based on the criterion of the American Diabetes Association
* being treated with oral antidiabetic medications
* able to speak and understand Mandarin
* able to walk without assistance
* have no regular exercise habit
* agree to join in a 12-week moderate-intensity exercise training after passing a graded exercise test.

Exclusion Criteria:

* receiving insulin therapy
* a history of cancer, end-stage renal disease with dialysis
* inability to participate in exercise training due to comorbid neurological and musculoskeletal conditions
* severe comorbidity or complications such as heart failure, autonomic neuropathy, and recent stroke within 6 months.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
exercise-induced glucose response | 12 weeks
  trend analysis of exercise-induced glucose response following a 12-week exercise training

SECONDARY OUTCOMES:
metabolic control/ trend of before-exercise blood glucose | 12 weeks
  trend analysis of before-exercise blood glucose following a 12-week exercise training
trend of post-exercise blood glucose | 12 weeks
  trend analysis of post-exercise blood glucose following a 12-week exercise training

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Huei Lin, PhD, Principal Investigator — Tri-Service General Hospital

IPD SHARING:
Plan to Share IPD: Undecided
After our research results were published. We will share our Study Protocol, Statistical Analysis Plan (SAP), and Clinical Study Report (CSR).

REFERENCES:
- [Result] Duclos M, Virally ML, Dejager S. Exercise in the management of type 2 diabetes mellitus: what are the benefits and how does it work? Phys Sportsmed. 2011 May;39(2):98-106. doi: 10.3810/psm.2011.05.1899. PMID 21673489
- [Result] Karjalainen JJ, Kiviniemi AM, Hautala AJ, Piira OP, Lepojarvi ES, Perkiomaki JS, Junttila MJ, Huikuri HV, Tulppo MP. Effects of physical activity and exercise training on cardiovascular risk in coronary artery disease patients with and without type 2 diabetes. Diabetes Care. 2015 Apr;38(4):706-15. doi: 10.2337/dc14-2216. Epub 2015 Jan 15. PMID 25592198
- [Result] Koivula RW, Tornberg AB, Franks PW. Exercise and diabetes-related cardiovascular disease: systematic review of published evidence from observational studies and clinical trials. Curr Diab Rep. 2013 Jun;13(3):372-80. doi: 10.1007/s11892-013-0373-0. PMID 23494754
- [Result] Rohling M, Herder C, Roden M, Stemper T, Mussig K. Effects of Long-Term Exercise Interventions on Glycaemic Control in Type 1 and Type 2 Diabetes: a Systematic Review. Exp Clin Endocrinol Diabetes. 2016 Sep;124(8):487-494. doi: 10.1055/s-0042-106293. Epub 2016 Jul 20. PMID 27437921
- [Result] Colberg SR, Sigal RJ, Fernhall B, Regensteiner JG, Blissmer BJ, Rubin RR, Chasan-Taber L, Albright AL, Braun B; American College of Sports Medicine; American Diabetes Association. Exercise and type 2 diabetes: the American College of Sports Medicine and the American Diabetes Association: joint position statement executive summary. Diabetes Care. 2010 Dec;33(12):2692-6. doi: 10.2337/dc10-1548. No abstract available. PMID 21115771
- [Result] Gulve EA. Exercise and glycemic control in diabetes: benefits, challenges, and adjustments to pharmacotherapy. Phys Ther. 2008 Nov;88(11):1297-321. doi: 10.2522/ptj.20080114. Epub 2008 Sep 18. PMID 18801852
- [Result] Way KL, Hackett DA, Baker MK, Johnson NA. The Effect of Regular Exercise on Insulin Sensitivity in Type 2 Diabetes Mellitus: A Systematic Review and Meta-Analysis. Diabetes Metab J. 2016 Aug;40(4):253-71. doi: 10.4093/dmj.2016.40.4.253. Epub 2016 Aug 2. PMID 27535644